CLINICAL TRIAL: NCT03725332
Title: The PATH Home Trial: A Comparative Effectiveness Study of Peripartum Opioid Use Disorder in Rural Kentucky
Acronym: PATH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wendy F Hansen (Other)
Responsible Party: Sponsor-Investigator, Wendy F Hansen, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 44929; MAT-2017C2-7842 (Other: Patients Centered Outcomes Research Institute)
Record Dates: First submitted 2018-10-29; First posted 2018-10-31 (Actual); Results first posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Neonatal Abstinence Syndrome
MeSH Terms: conditions — Neonatal Abstinence Syndrome | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine Education (Experimental): This is a stratified cluster non-inferiority randomized controlled trial with randomization of participating clusters into a 'telemedicine' or 'group care' arm. Sites will be stratified into 'high volume' (>500 deliveries/year) and 'low volume' (<500 deliveries per year). Randomization will be within each strata. Patients attending sites randomized to telemedicine will be recruited by research staff.
  Interventions: Behavioral: Telemedicine
- Group Care Education (Active Comparator): This is a stratified cluster non-inferiority randomized controlled trial with randomization of participating clusters into a 'telemedicine' or 'group care' arm. Sites will be stratified into 'high volume' (>500 deliveries/year) and 'low volume' (<500 deliveries per year). Randomization will be within each strata. Patients attending sites randomized to group care will be recruited by research staff.
  Interventions: Behavioral: Group Care

INTERVENTIONS:
Behavioral: Telemedicine — Patients enrolled at sites randomized to telemedicine will receive a standardized, rotating patient education curriculum through consultations with substance use counselor or perinatal nurse facilitator. Consultations will occur twice a month until 8 weeks post-partum and will then continue monthly until 6 months postpartum. Rotating topics include: 1) Treatment Options for Opioid Use Disorder, 2) Smoking Cessation, 3) Relapse Prevention Education, 4) NAS Reduction Education, 5) Breast Feeding Support/Education, 6) Domestic Violence Education, 7) Postpartum Depression, and 8) Birth Control/Family Planning.
  Arms: Telemedicine Education
Behavioral: Group Care — Patients enrolled at sites randomized to group care will receive a standardized, rotating patient education curriculum delivered in small groups led by a perinatal nurse facilitator or substance use counselor, with a peer support specialist. Small group care meetings will occur twice a month until 8 weeks post-partum and will then continue monthly until 6 months post-partum. Rotating topics include: 1) Treatment Options for Opioid Use Disorder, 2) Smoking Cessation, 3) Relapse Prevention Education, 4) NAS Reduction Education, 5) Breast Feeding Support/Education, 6) Domestic Violence Education, 7) Postpartum Depression, and 8) Birth Control/Family Planning.
  Arms: Group Care Education

SUMMARY:
Perinatal opioid use disorder (OUD) is a major health concern in the U.S. with significant impact on mothers, infants, and communities. Investigators at the University of Kentucky/UK HealthCare (UK) have developed a comprehensive clinical care model for perinatal OUD (known as UK-PATHways) that has demonstrated success in maternal and neonatal outcomes. The overreaching goals of the proposed project are to: 1) expand the reach of this successful clinical program to rural communities thereby improving access to integrated MAT prenatal care, 2) to reduce the impact of perinatal OUD in underserved rural areas of our state, and 3) to compare the relative effectiveness methods of delivery active elements of the UK-PATHways program for rural implementation (local group-support vs. telemedicine).

DETAILED DESCRIPTION:
The UK-PATHways program preliminary successes during the first three years are clear: enrolled mothers (n>200) have reduced relapse, increased treatment compliance, and improved neonatal outcomes when compared to non-enrolled OUD mothers. However, at this time, UK-PATHways is only available at the main healthcare campus in Lexington, KY. Many eligible patients reside great distances from our clinical home and some current patients travel hours to access this valuable resource. While Medication Assisted Therapy (MAT) has become increasingly available in our region, many of the components of the UK-PATHways program are not readily accessible in rural Central and Eastern Kentucky and the quality of programming with MAT treatment is not standardized in these locations. Furthermore, rural patients continue to face challenges related to stigma of their OUD and transportation difficulties if they desire more comprehensive services. The proposed study will evaluate the introduction of essential components of the UK-PATHways program into rural communities and identify the optimal intervention strategies for expansion of services and to improve the treatment of OUD for rural patients. Specific aims include the following: Aim 1) Conduct a randomized cluster trial using a 'hub and spoke' study design, comparing two delivery modes (local GROUP care vs TELEMEDICINE) for the delivery of a UK-PATHways based patient education curriculum at participating rural regional sites. Each regional site will be randomized to support one of two study arms: 1) Prenatal group care led by a perinatal nurse facilitator or substance use counselor with a peer support specialist (GROUP arm); or, 2) Telemedicine consultation with substance use counselor or perinatal nurse facilitator based at the 'hub' site (TELEMEDICINE arm); and Aim 2) Evaluate the relative effectiveness of each study arm on primary and secondary maternal and neonatal outcomes as compared to the established UK-PATHways program (UK PATHways: Hub) at the University of Kentucky.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at 6 to 32 weeks' gestational age
* History of Opioid Use Disorder
* Receiving Medication Assisted Therapy (buprenorphine products or methadone)
* Obtaining prenatal care at one of eleven study sites located throughout Central and Eastern Kentucky

Exclusion Criteria:

-

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 269 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Hansen, MD, Principal Investigator — University of Kentucky, Department of OB-GYN, Division of Maternal Fetal Medicine
Locations (11):
- United States (11):
  - Karen's Place Maternity Center, Ashland, Kentucky
  - The Medical Center, Bowling Green, Kentucky
  - Grace Health Women's Care, Corbin, Kentucky
  - BrightView, Georgetown, Kentucky
  - University of Kentucky Women's Health OB-GYN, Georgetown, Kentucky
  - Primary Care Centers of Eastern Kentucky, Hazard, Kentucky
  - OB/GYN & Women's Health University of Louisville, Louisville, Kentucky
  - ARH Women's and Family Health Center - Middlesboro, Middlesboro, Kentucky
  - University of Kentucky Morehead Women's Healthcare, Morehead, Kentucky
  - Frontier Behavioral Health Centers, Prestonsburg, Kentucky
  - ARH Women's and Family Health Center - Tug Valley, South Williamson, Kentucky

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD at this time

RESULTS

PARTICIPANT FLOW:
Recruitment Details: On 8/30/2019 study design was changed to a non-inferiority and recruitment to 533. Unable to meet 533 within the time frame and budget allotted, 4 secondary outcomes were powered: Urine drug screen at delivery, number of interventions, prenatal visits and MAT visits attended. On 8/2022, recruitment target changed to 256-80 participants in telemedicine, and 176 in group. Final enrollment was 269. Enrollment occurred between 3/13/19-10/16/23 at 13 sites.
Pre-assignment Details: Randomization to Group or Telemedicine was at the site level. All enrollments were predetermined by the site which the women enrolled. There was no period between enrollment and assignment. Enrollment and assignment occurred simultaneously. Wash out- periods and Run-in periods are not applicable to this study
Units Other Than Participants: study sites
Period: Overall Study
Arm/Group | Telemedicine Education | Group Care Education
Started | 82; 6 study sites | 187; 7 study sites
At Delivery | 79; 6 study sites | 175; 7 study sites
At 4 Weeks Postpartum | 33; 6 study sites | 70; 7 study sites
At 3 Months Postpartum | 37; 6 study sites | 58; 7 study sites
Completed | 33; 6 study sites | 49; 7 study sites
Not Completed | 49; 0 study sites | 138; 0 study sites
Not completed — Adverse Event | 5 | 10
Not completed — Death | 1 | 3
Not completed — Lost to Follow-up | 43 | 122
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Duplicate enrollment | 0 | 1
Not completed — Did not consent | 0 | 1

BASELINE CHARACTERISTICS:
Population: Three Group Arm participants were not assessed due to administrative errors.
Groups:
- Total: Total of all reporting groups
Arm/Group | Telemedicine Education | Group Care Education | Total
Number analyzed (Participants) | 82 | 184 | 266
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 82 | 184 | 266
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.4 (4.8) | 30.1 (5.4) | 30.2 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 184 | 266
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 78 | 182 | 260
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 78 | 181 | 259
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 82 | 184 | 266

OUTCOME MEASURES:

1. Primary Outcome: Percent of Infants Diagnosed With Neonatal Abstinence Syndrome (NAS) Requiring Medication Treatment
Description: Medical records will be reviewed post-partum for treatment for NAS. Diagnosis of NAS will be made within 10 days of birth and treatment started based on standard of care. Data will be presented as the percent of infants born requiring therapy in each group.
Time Frame: up to 10 days postpartum
Population: Number of participants (infants) available for data analysis per protocol
Measure: Number; unit: % infants requiring medication for NAS
Arm/Group | Telemedicine Education | Group Care Education
Number analyzed (Participants) | 80 | 177
% infants requiring medication for NAS | 24.1 | 33.3

2. Secondary Outcome: Number of Inappropriate Maternal Drug Screens at Delivery
Description: Maternal urine drug screen (UDS) will be collected at the time of hospital admission for delivery for each participant. A urine drug screen is considered inappropriate when the presence of an illicit drug that is not prescribed for the participant is detected or the prescribed medication for opioid use disorder is not detected. The actual number of inappropriate maternal drug screens will be calculated. Results will be compared between Arms: Telemedicine and Group
Time Frame: Up to 10 days post-partum
Population: Participants available for data analysis per protocol
Measure: Number; unit: # of inappropriate maternal drug screens
Arm/Group | Telemedicine Education | Group Care Education
Number analyzed (Participants) | 63 | 164
# of inappropriate maternal drug screens | 12 | 29

3. Secondary Outcome: Prenatal Engagement With Percent of Program Education Sessions Attended
Description: Engagement with PATHHome is measured by the number of counseling/education sessions (groups or telemedicine) attended by each participant. Results will be compared between Arms and expressed as percent of interventions attended by participants.
Time Frame: Up to delivery, an average of 19 weeks
Population: Number of participants available for data analysis per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Telemedicine Education | Group Care Education
Number analyzed (Participants) | 79 | 175
Participants
  No intervention attended | 12 | 36
  5-50% interventions attended | 26 | 62
  51-100% interventions attended | 41 | 77

4. Secondary Outcome: Prenatal Engagement With MAT Provider
Description: Engagement with MAT provider is measured by the average number of visits attended by each participant with their MAT provider.
Time Frame: Up to delivery, an average of 19 weeks
Population: Number of participants available for data analysis per protocol
Measure: Mean (Standard Error); unit: Visits
Arm/Group | Telemedicine Education | Group Care Education
Number analyzed (Participants) | 82 | 184
Visits | 12.0 (1.70) | 8.40 (0.65)

5. Secondary Outcome: Prenatal Engagement in Prenatal Care
Description: Engagement with Prenatal Care is considered by gestational age of entry. The number of prenatal visits is expressed as a percentage of prenatal visits attended with a denominator of prenatal visits scheduled. The data is provided by patient report and confirmed by medical record review when possible. Results will be compared between Arms. Categories reported are no prenatal visits, 5-50%, 51-100%.
Time Frame: Up to delivery, an average of 19 weeks
Population: Number of participants available for data analysis per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Telemedicine Education | Group Care Education
Number analyzed (Participants) | 79 | 175
Participants
  No prenatal care visits | 4 | 11
  5-50% prenatal care visits | 16 | 35
  51-100% prenatal care visits | 59 | 129

6. Secondary Outcome: Participants With Cigarette Dependency Over Time
Description: Participants will complete the Fagerstrom Test for Cigarette Dependence 4 times during the course of the study: Intake, 28-32 weeks, 3 months postpartum and 6 months postpartum (combined total time of observation is up to 60 weeks). This is a 7-question survey with each question scored on a scale of zero to 3 and totaled. Scores greater than 8 are considered high dependency, scores of 5-7 are considered moderately dependent, scores of 3-4 are low to moderate dependence and scores of 1-2 are low dependence. Data will be presented as the number of participants with cigarette dependency over time compared between groups.
Time Frame: Up to 60 weeks
Population: Number of participants available for data analysis per protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Telemedicine Education | Group Care Education
Number analyzed (Participants) | 82 | 184
Participants
  Intake: number analyzed (Participants) | 75 | 171
  Intake: 0: None; Former or never smoker | 14 | 42
  Intake: 1-2: Low dependency | 7 | 20
  Intake: 3-4: low- moderate dependency | 15 | 28
  Intake: 5-7: Moderate dependency | 27 | 64
  Intake: 8-10: High dependency | 12 | 17
  28-32weeks: number analyzed (Participants) | 42 | 89
  28-32weeks: 0: None; Former or never smoker | 10 | 23
  28-32weeks: 1-2: Low dependency | 4 | 10
  28-32weeks: 3-4: low- moderate dependency | 8 | 23
  28-32weeks: 5-7: Moderate dependency | 12 | 29
  28-32weeks: 8-10: High dependency | 8 | 4
  3 months postpartum: number analyzed (Participants) | 31 | 49
  3 months postpartum: 0: None; Former or never smoker | 5 | 16
  3 months postpartum: 1-2: Low dependency | 2 | 9
  3 months postpartum: 3-4: low- moderate dependency | 4 | 7
  3 months postpartum: 5-7: Moderate dependency | 12 | 13
  3 months postpartum: 8-10: High dependency | 8 | 4
  6 months postpartum: number analyzed (Participants) | 26 | 39
  6 months postpartum: 0: None; Former or never smoker | 4 | 17
  6 months postpartum: 1-2: Low dependency | 3 | 6
  6 months postpartum: 3-4: low- moderate dependency | 6 | 7
  6 months postpartum: 5-7: Moderate dependency | 8 | 7
  6 months postpartum: 8-10: High dependency | 5 | 2

7. Secondary Outcome: Participants With Maternal Anxiety Over Time
Description: Participants will complete the Generalized Anxiety Disorder survey at their intake visit, at 28-32 weeks, 3 months postpartum and 6 months postpartum (combined total time of observation is up to 60 weeks). The survey consists of 7 questions probing the participants burden of anxiety. Each question is scored from 0 to 3, with 3 representing the most severe state. A total score of 1-4 indicates minimal anxiety, 5-14 indicates moderate anxiety, and 15-21 indicates severe anxiety. Data will be presented as the number of participants with anxiety over time compared between groups.
Time Frame: Up to 60 weeks
Population: Number of participants available for data analysis per protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Telemedicine Education | Group Care Education
Number analyzed (Participants) | 82 | 184
Participants
  Intake: number analyzed (Participants) | 77 | 171
  Intake: '0': No anxiety | 7 | 23
  Intake: 1-4: Minimal anxiety | 16 | 50
  Intake: 5-14 Moderate anxiety | 43 | 78
  Intake: 15-21 Severe anxiety | 11 | 20
  28-32 weeks: number analyzed (Participants) | 47 | 91
  28-32 weeks: '0': No anxiety | 5 | 23
  28-32 weeks: 1-4: Minimal anxiety | 11 | 27
  28-32 weeks: 5-14 Moderate anxiety | 26 | 34
  28-32 weeks: 15-21 Severe anxiety | 5 | 7
  3 months postpartum: number analyzed (Participants) | 31 | 49
  3 months postpartum: '0': No anxiety | 6 | 11
  3 months postpartum: 1-4: Minimal anxiety | 10 | 13
  3 months postpartum: 5-14 Moderate anxiety | 15 | 20
  3 months postpartum: 15-21 Severe anxiety | 0 | 5
  6 months postpartum: number analyzed (Participants) | 26 | 39
  6 months postpartum: '0': No anxiety | 6 | 10
  6 months postpartum: 1-4: Minimal anxiety | 7 | 10
  6 months postpartum: 5-14 Moderate anxiety | 11 | 18
  6 months postpartum: 15-21 Severe anxiety | 2 | 1

8. Secondary Outcome: Participants With Maternal Depression Over Time
Description: Participants will complete the Edinburgh Depression Scale at 4 times during the study: Intake visit, at 28-32 weeks, 3 months postpartum and 6 months postpartum (combined total time of observation is up to 60 weeks). The survey consists of 10 questions. Each question is scored between 0-3. An answer of 3 represents a more severe state. A total score of 1-8 falls within a normal range, a score is 9-10 is at risk for depression and a score of 11 or more indicates depression. In general, the higher the score, the more severe the depression. Data will be presented as the number of participants with depression over time compared between groups.
Time Frame: Up to 60 weeks
Population: Number of participants available for data analysis per protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Telemedicine Education | Group Care Education
Number analyzed (Participants) | 82 | 184
Participants
  Intake: number analyzed (Participants) | 78 | 167
  Intake: 1-8: Normal | 24 | 60
  Intake: 9-10: At risk for depression | 8 | 19
  Intake: 11-29: Depression | 46 | 88
  28-32 weeks: number analyzed (Participants) | 46 | 85
  28-32 weeks: 1-8: Normal | 21 | 38
  28-32 weeks: 9-10: At risk for depression | 5 | 10
  28-32 weeks: 11-29: Depression | 20 | 37
  3 months postpartum: number analyzed (Participants) | 31 | 45
  3 months postpartum: 1-8: Normal | 20 | 19
  3 months postpartum: 9-10: At risk for depression | 2 | 10
  3 months postpartum: 11-29: Depression | 9 | 16
  6 months postpartum: number analyzed (Participants) | 23 | 35
  6 months postpartum: 1-8: Normal | 13 | 15
  6 months postpartum: 9-10: At risk for depression | 1 | 7
  6 months postpartum: 11-29: Depression | 9 | 13

9. Secondary Outcome: Participant Quality of Life
Description: WHO-Quality of Life Survey (WHOQoL) will be administered to patients at 28-32 weeks gestation. WHOQoL is a 26 question self administered survey. Each question falls within 1 of 4 "domains": physical health, psychological health, social relationships, environment. For purposes of reporting, we are using the first question, "How would you rate your quality of life?" on a scale of 1-5, with 1 being very poor quality, 2 poor quality, 3 neither poor nor good, 4 good quality, 5 very good quality.
Time Frame: 28-32 weeks gestation
Population: Number of participants available for data analysis per protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Telemedicine Education | Group Care Education
Number analyzed (Participants) | 46 | 91
Participants
  Very Good quality of life | 18 | 29
  Good quality of life | 26 | 55
  Neither poor nor good quality of life | 2 | 6
  Poor quality of life | 0 | 1
  Very poor quality of life | 0 | 0

10. Secondary Outcome: Severity of Opioid Use Disorder
Description: Participants will complete a Diagnostic and Statistical Manual of Mental Disorders-5-TR, Addiction Severity Scale to assess their opioid dependency at the intake visit (between 6-32 weeks). The survey asks 11 questions. Each question asks about symptoms related to opioid use disorder and are answered in a yes/no format. A mild substance use disorder is diagnosed with 2-3 symptoms, moderate with 4-5 symptoms, and severe is 6 or more symptoms. Data will be presented as the number of participants in each category.
Time Frame: Intake visit (between 6-32 weeks gestation)
Population: Number of participants available for data analysis per protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Telemedicine Education | Group Care Education
Number analyzed (Participants) | 82 | 184
Participants
  0-1: None/Minimal | 41 | 65
  2-3: Mild | 8 | 25
  4-5: Moderate | 7 | 15
  6-11: Severe | 22 | 63

11. Secondary Outcome: Incidence of Hospitalization for Opioid Related Issues During the Study Period
Description: Hospitalizations for opioid related issues were determined by two main methods. Participants were assessed for hospitalization at each intervention visit. Interventions occurred every two weeks until 8 weeks postpartum, then monthly through 6 months. Secondly, hospitalizations were determined and confirmed through medical record review when possible. Data will be presented as number of hospitalizations in each arm.
Time Frame: up to 60 weeks
Population: Number of participants available for data analysis per protocol
Measure: Number; unit: Numbe of hospitalizations
Arm/Group | Telemedicine Education | Group Care Education
Number analyzed (Participants) | 82 | 184
Numbe of hospitalizations | 2 | 4

12. Secondary Outcome: Change in Physical Condition of Infant Post-delivery by Apgar Score
Description: Infant physical condition at birth will be assessed using the Apgar score at 1 minute and 5 minutes after birth. The Apgar score consists of 5 criteria: Appearance (skin color), pulse, grimace (reflex irritability), activity (muscle tone), respiration. Each criteria is scored 0-2. Scores are summed to evaluate a newborns health. A score of 8-10 is considered normal. A score less than 8 requires medical support. The lower the score, the more severely affected the newborn. Data will be presented as the change in Apgar score over time compared between groups.
Time Frame: Up to five minutes
Population: Telemedicine arm had one set of twins; Group arm had two sets of twins. Number of participants available for data analysis per protocol
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Telemedicine Education | Group Care Education
Number analyzed (Participants) | 75 | 169
score on a scale
  1 minute after birth | 7.89 (0.14) | 7.94 (0.11)
  5 minutes after birth | 8.61 (0.10) | 8.76 (0.05)

13. Secondary Outcome: Incidence of Pediatric Emergency Room (ER) Visits
Description: Pediatric emergency room visits will be determined by both in person reporting during a postpartum intervention and by medical record review. Time span starts at discharge from the hospital (after birth) to 6 months postpartum. Data will be presented as the total number of pediarric ER visits compared between groups
Time Frame: birth-six months
Population: Number of infants available for data analysis per protocol
Measure: Number; unit: Number of infants
Arm/Group | Telemedicine Education | Group Care Education
Number analyzed (Participants) | 75 | 171
Number of infants | 10 | 11

14. Secondary Outcome: Adherence to a Vaccine Schedule
Description: Adherence to a vaccine schedule will be determined by both in person reporting during a postpartum intervention and by medical record review when possible. Participants will be asked at their 3 and 6-month postpartum visit; "Is your infant up to date on vaccines?". Data will be presented as the total number of infants compliant on their vaccines and compared between groups.
Time Frame: Infant 3 months and 6 months of age
Population: Number of infants available for data analysis per protocol
Measure: Number; unit: Number of infants
Arm/Group | Telemedicine Education | Group Care Education
Number analyzed (Participants) | 75 | 171
Number of infants
  Infant 3 months of age | 27 | 45
  Infant 6 months of age | 22 | 39

15. Secondary Outcome: Engagement With Pediatric Care
Description: Engagement with pediatric care will be determined by both in person reporting during a postpartum intervention and by medical record review when possible. Participants will be asked at their 3 and 6-month postpartum visit; "Does your baby regularly see a pediatrician?". Data will be presented as the total number of infants engaged in pediatric care and compared between groups.
Time Frame: Infant 3 month and 6 months of life
Population: Number of infants available for data analysis per protocol
Measure: Number; unit: Number of infants adhering
Arm/Group | Telemedicine Education | Group Care Education
Number analyzed (Participants) | 75 | 171
Number of infants adhering
  Infant 3 months of age | 30 | 49
  Infant 6 months of age | 26 | 42

16. Secondary Outcome: Infant Gross Motor Development
Description: The Ages & Stages Questionnaires®, Third Edition (ASQ®-3) was completed by the participant at the 3-month postpartum intervention. The survey collects infant milestones in five domains: communication, gross motor, fine motor, problem-solving, and personal/social. The developmental instrument is 38 items and scored by the research staff. For purposes of reporting, we are utilizing the gross motor domain subsection score only. This domain includes 6 questions. Scores are calculated at 0, 5, or 10 per question. The highest score is 60- the lowest score would be 0. The higher the score the better. For a score greater than 41 development is considered to be on schedule. If the score falls between 38-41- targeted learning activities and monitoring is recommended. If the score falls below 38, concern for lagging infant motor development and further assessment with a professional is recommended. Scores will be presented as the mean +/- standard error compared between group
Time Frame: Infant at 3 months of age
Population: Number of participants available for data analysis per protocol
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Telemedicine Education | Group Care Education
Number analyzed (Participants) | 75 | 171
score on a scale | 53.10 (1.52) | 55.22 (0.88)

17. Secondary Outcome: Infant Gross Motor Development
Description: The Ages & Stages Questionnaires®, Third Edition (ASQ®-3) was completed by the participant at the 6-month postpartum intervention. The survey collects infant milestones in five domains: communication, gross motor, fine motor, problem-solving, and personal/social. The Ages and Stages 6-month survey instrument is 38 items and scored by the research staff. For purposes of reporting, we are utilizing the gross motor domain score only. This domain includes 6 questions, scores are calculated at 0, 5, or 10 per question and a score below 22 is concerning for lagging infant motor development. Scores will be presented as the mean +/- standard error compared between groups.
Time Frame: Infant at 6 months of age
Population: Number of infants available for data analysis per protocol
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Telemedicine Education | Group Care Education
Number analyzed (Participants) | 75 | 171
score on a scale | 50.40 (2.71) | 48.71 (1.41)

18. Secondary Outcome: Incidence of Relapse
Description: Relapse was defined as the use of any illicit substance or misuse of prescribed medications including medication for opioid use disorder. Incidence of relapse was determined by two main methods. Participants were assessed for relapse at each intervention visit. Interventions occurred every two weeks until 8 weeks postpartum, then monthly through 6 months. Secondly, relapses were determined and confirmed through medical record review, including inappropriate urine drug screens, when possible. Data will be presented in 2 categories: Relapse with opioids and relapse with other substances. The number of relapses is not equal to the number of participants as a single participant may have more than one relapse or polysubstance relapse. Data will be presented as the total number of relapses and compared between groups.
Time Frame: Up to 60 weeks
Population: Number of participants available for data analysis per protocol
Measure: Number; unit: Number of relapses
Arm/Group | Telemedicine Education | Group Care Education
Number analyzed (Participants) | 82 | 184
Number of relapses
  Relapse with opioids | 10 | 29
  Relapse with other substances | 37 | 188

19. Secondary Outcome: Incidence of Opioid Overdose
Description: The incidence of opioid overdose was determined by two main methods. Participants were assessed for overdose at each intervention visit. Interventions occurred every two weeks until 8 weeks postpartum, then monthly through 6 months. Secondly, overdoses were determined and confirmed through medical record review when possible. Data will be presented as number of overdoses in each arm.
Time Frame: Up to 60 weeks
Population: Number of participants available for data analysis per protocol
Measure: Number; unit: Number of opioid overdoses
Arm/Group | Telemedicine Education | Group Care Education
Number analyzed (Participants) | 82 | 184
Number of opioid overdoses | 0 | 4

20. Other Pre Specified Outcome: Change in Employment Status
Description: Participants will be asked about employment status during their intake visit, at 28 weeks gestational age, 3 months postpartum and 6 months postpartum (combined total time of observation is up to 60 weeks). Participants will answer "yes" or "no" regarding their employment status. Data will be presented as the change in employment status between groups.
Time Frame: Up to 60 weeks
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Change in Household Size
Description: Participants will be asked to indicate the total number of people sharing their living space during the intake visit, and 6 months postpartum (combined total time of observation is up to 38 weeks). Data will be presented as the change in dwelling occupancy over time compared between groups.
Time Frame: up to 38 weeks
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Acceptance of Long-term Contraception
Description: Participants will be offered long-acting reversible contraception. Data will be presented as the number of participants per group accepting long term contraception.
Time Frame: Up to 6 months postpartum
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From enrollment (between 6-32 weeks pregnant) until infant is 6 months old.
Description: Definition of adverse event and serious adverse event matches the clinicaltrials.gov definitions. Infant adverse events were not part of the research plan. Adverse events only collected on mothers. Three Group Arm participants were not assessed due to administrative errors.
Arm/Group | Telemedicine Education | Group Care Education
All-Cause Mortality (participants affected / at risk) | 1/82 | 3/184
Serious Adverse Events (participants affected / at risk) | 20/82 | 46/184
Other Adverse Events (participants affected / at risk) | 72/82 | 166/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telemedicine Education (N=82) | Group Care Education (N=184)
Preterm labor (Pregnancy, puerperium and perinatal conditions) | 5 (7) | 5 (5)
Non-reactive NST/Elevated dopplers (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 4 (4)
Placental abruption (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 4 (6)
Preeclampsia (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 2 (2)
IUGR (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
PPROM (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Hydrops fetalis (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Spontaneous abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Vaginal bleeding (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
C-section wound dehiscence (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Hemorrhagic shock (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Opioid overdose (Psychiatric disorders) | 0 (0) | 3 (3)
Overdose - unknown substance (Psychiatric disorders) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0) — Due to IV drug use
Opioid withdrawal (Psychiatric disorders) | 1 (1) | 0 (0)
Severe OUD (Psychiatric disorders) | 0 (0) | 1 (1)
Diffuse anoxic brain injury (Nervous system disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Viral Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 1 (1)
C-section wound infection (Infections and infestations) | 0 (0) | 1 (1)
Acute Hep C superimposed on chronic (Infections and infestations) | 0 (0) | 1 (1)
Acute Exacerbation of Chronic Pancreatitis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Trauma/Injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Acute hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Infant death (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1)
Transaminitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Psychiatric (Psychiatric disorders) | 1 (1) | 0 (0)
Hemorrhage (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Acute cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Acute pyelonephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Abdominal Cramping/Pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Acute appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Right mastectomy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1)
Renal Agenesis of fetus (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telemedicine Education (N=82) | Group Care Education (N=184)
Respiratory (Infections and infestations) | 11 (15) | 9 (10)
IUGR (Pregnancy, puerperium and perinatal conditions) | 13 (13) | 23 (23)
Relapse THC (Psychiatric disorders) | 9 (11) | 30 (36)
Urinary (Renal and urinary disorders) | 6 (11) | 24 (26) — infections
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 11 (11) | 10 (10)
MAT misuse (Psychiatric disorders) | 10 (12) | 28 (31)
Relapse opioids (Psychiatric disorders) | 9 (10) | 18 (29)
Relapse amphetamines (Psychiatric disorders) | 6 (9) | 36 (46)
Preterm labor (Pregnancy, puerperium and perinatal conditions) | 7 (9) | 19 (25)
Fetal distress, non-reactive NST/Elevated Dopplers, non-reassuring BPP (Pregnancy, puerperium and perinatal conditions) | 8 (9) | 17 (17)
Pain (General disorders) | 4 (9) | 10 (12) — abdomen
Dental (Gastrointestinal disorders) | 8 (9) | 10 (10)
Relapse benzodiazepines (Psychiatric disorders) | 5 (8) | 17 (18)
Gestational Hypertension (Pregnancy, puerperium and perinatal conditions) | 6 (7) | 19 (21)
Relapse gabapentin (Psychiatric disorders) | 5 (6) | 22 (38)
STI (Infections and infestations) | 5 (6) | 11 (19)
COVID (Infections and infestations) | 6 (6) | 15 (15)
Illicit Suboxone Use (Psychiatric disorders) | 4 (4) | 20 (30)
Postpartum Depression (Psychiatric disorders) | 4 (4) | 14 (14)
ENT (Ear and labyrinth disorders) | 7 (7) | 9 (10)

LIMITATIONS AND CAVEATS:
The study is NOT powered for the primary outcome NAS, but is powered for 4 major secondary outcomes- maternal urine drug screen at delivery, and the number of education/interventions, prenatal care and MAT visits attended Protocols for NAS treatment differ greatly between hospitals and potentially effect the start and the type of medication treatment Complex data collection relying on frequent participant interviews and medical records Patients would be LTFU and then return to the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-22): https://cdn.clinicaltrials.gov/large-docs/32/NCT03725332/Prot_SAP_000.pdf